CLINICAL TRIAL: NCT06664190
Title: Study on Preoperative Imaging for Precise Prediction of Surgical Difficulty, Efficacy, and Risks in Pituitary Adenoma Surgeries
Brief Title: Pre-operative Surgical Difficulty Stratification Using Predicted Tumor Perfusion and Consistency
Status: Active, not recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Professor, Huashan Hospital
Other Study IDs: KY2022-709
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Advanced sequences, such as arterial spin labeling (ASL) and diffusion-weighted imaging (DWI) — Advanced sequences, such as arterial spin labeling (ASL) and diffusion-weighted imaging (DWI)

SUMMARY:
Pituitary adenomas (PAs) are among the most prevalent lesions of the sella turcica, accounting for 10%-25% of all intracranial neoplasms. Pituitary macroadenomas (PMAs) are defined with a maximum diameter of over 1 cm. Tumor characteristics are key factors influencing surgical effectiveness and complications of PMAs, with tumor perfusion and consistency identified as major predictive factors in literature. Conventional sequences provide limited information for predicting the perfusion and consistency of pituitary adenomas. Advanced sequences offer additional insights. However, the efficacy of combining radiomic features from multiparametric sequences, incorporating both conventional and advanced sequences, has not yet been proved.

We aim to develop machine learning models that combines radiomic features developed from both conventional and advanced sequences to predict the perfusion and consistency of PMAs. Furthermore, we aim to demonstrate the clinically applicability of these models by constructing a MR-PIT stratification (Multiparametric Radiomic derived and tumor Perfusion and consIsTency based surgical difficulty stratification), which correlated with the surgical strategy and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients with tumor more than 2.5 cm of maximal diameter in the coronal plane
* Functional and non-functional pituitary tumors

Exclusion Criteria:

* incomplete image data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients histologically diagnosed with pituitary adenomas and who had undergone surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Extent of resection | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
Severe postoperative complications | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No